CLINICAL TRIAL: NCT01547715
Title: A Phase 3, Multi-center, Open-label Study to Evaluate Immunogenicity and Safety of Novartis Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) in Healthy Subjects From 2 to 75 Years of Age in India.
Brief Title: Immunogenicity and Safety of Meningococcal ACWY Conjugate Vaccine in Healthy Subjects From 2 to 75 Years of Age in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V59_43
Record Dates: First submitted 2012-02-23; First posted 2012-03-08 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Bacterial Meningitis
Keywords: Meningococcal,; ACWY,; bacterial meningitis,; conjugate vaccine,; healthy, children,; adolescents,; adults,; India
MeSH Terms: conditions — Meningitis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MenACWY - 2 - 10 Years old (Experimental): Subjects between 2 and 10 years of age who received one injection of Meningococcal ACWY conjugate vaccine -CRM vaccine on day 1.
  Interventions: Biological: Meningococcal ACWY conjugate vaccine
- MenACWY - 11 - 18 Years old (Experimental): Subjects between 11 and 18 years of age who received one injection of Meningococcal ACWY conjugate vaccine-CRM vaccine on day 1.
  Interventions: Biological: Meningococcal ACWY conjugate vaccine
- MenACWY - 19 - 75 Years old (Experimental): Subjects between 11 and 18 years of age who received one injection of Meningococcal ACWY conjugate vaccine-CRM vaccine on day 1.
  Interventions: Biological: Meningococcal ACWY conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal ACWY conjugate vaccine — All subjects received a single dose of Meningococcal ACWY conjugate vaccine

SUMMARY:
This study will evaluate the immunogenicity of a single injection of Novartis Meningococcal ACWY conjugate vaccine in healthy subjects from the age of 2 years and above in India.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrollment in this study are those:

1. who are of any gender, from the age of 2 to 75 years at the time of visit 1, and to whom the nature of the study has been explained and:

   * the parent/legal representative has provided written informed consent (greater than or equal to 2 - less than 18 years of age).
   * have provided written assent (greater than or equal to 7-less than or equal to 18 years)
   * have provided written informed consent (greater than or equal to 18 to 75 years of age).
2. who the investigator believes that they or their parents/legal representatives can and will comply with the requirements of the protocol (e.g., completion of the Diary Card, return for follow-up visit).
3. who are in good health as determined by medical history, physical exam, clinical judgment of the investigator
4. who have a negative urine pregnancy test for female subjects of childbearing potential.

Exclusion Criteria:

Individuals not eligible to be enrolled in the study are those:

1. who are unwilling or unable to give written informed assent or consent to participate in the study.
2. who are perceived to be unreliable or unavailable for the duration of the study period.
3. who had a previous or suspected disease caused by N. meningitidis.
4. who had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis infection within 60 days prior to enrollment.
5. who have previously been immunized with a meningococcal vaccine.
6. who have received any investigational or non-registered product (drug or vaccine)within 28 days prior to enrollment or who expect to receive an investigational drug or vaccine prior to the completion of the study.
7. who have received any vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who are planning to receive any vaccine within 30 days from the study vaccines. (Exception: Influenza vaccine may be administered up to 15 days prior to study vaccination and at least 15 days after study vaccination)
8. who have experienced within the 7 days prior to enrollment significant acute infection (for example requiring systemic antibiotic treatment or antiviral therapy) or have experienced fever (defined as body temperature greater than or equal to 38°C) within 3 days prior to enrollment.
9. who have any serious acute, chronic or progressive disease (e.g., any history of neoplasm, cancer, diabetes, cardiac disease, autoimmune disease, HIV infection or AIDS, or blood dyscrasias, with signs of cardiac or renal failure or severe malnutrition).
10. who have epilepsy or any progressive neurological disease.
11. who have a history of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine components.
12. who have a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from (for example):

    * receipt of immunosuppressive therapy within 28 days prior to enrollment (any systemic corticosteroid administered for more than 5 days, or in a daily dose greater than 1 mg/kg/day prednisone or equivalent during any of 28 days prior to enrollment, or cancer chemotherapy)
    * receipt of immunostimulants
    * receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 90 days prior to enrollment and for the full length of the study.
13. who are known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
14. who have any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Lalwani, Principal Investigator — Bharati Hospital and Research Center; Dr. Nitya Gogtay, Principal Investigator — Seth GS Medical College and KEM Hospital; Dr. A Amaresh, Principal Investigator — Niloufer Hospital, Hyderabad; Dr. Sharad Agarkhedkar, Principal Investigator — Padmasree Dr. D.Y.patil Medical College, Hospital & Research Center
Locations (4):
- India (4):
  - Osmania Medical College Ethics Commitee, Niloufer Hospital, Hyderabad, Andrapradesh
  - Bharati Vidyapeeth University Institutional Ethics Commitee, Katraj, Dhankawadi
  - Seth GS Medical College and KEM Hospital, Mumbai, Maharashtra
  - Padmasree Dr. D.Y Patil medical College, Pune, Maharashtra

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 3 study sites.
Pre-assignment Details: All the enrolled subjects were included in the trial.
Groups:
- 2 - 10 Years: Subjects between 2 and 10 years of age received one injection of MenACWY -CRM vaccine on day 1.
- 11 - 18 Years: Subjects between 11 and 18 years of age received one injection of MenACWY -CRM vaccine on day 1.
- 19 - 75 Years: Subjects between 19 and 75 years of age received one injection of MenACWY -CRM vaccine on day 1.
Period: Overall Study
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years
Started | 60 | 60 | 60
Completed | 60 | 60 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 5.77 (2.5) | 14.03 (1.931) | 32.67 (12.297) | 17.49 (13.432)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 33 | 33 | 21 | 87
  MALE | 27 | 27 | 39 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Human Serum Bactericidal Assay (hSBA) Seroresponse Against N.Meningitidis Serogroup A.
Description: The immunogenicity of a single injection of MenACWY-CRM vaccine is assessed in terms of percentage of subjects with hSBA seroresponse directed against N.meningitidis serogroup A. Seroresponse is defined as:
  * For subjects with a pre-vaccination hSBA titer <1:4, a postvaccination hSBA titer≥1:8
  * For subjects with a pre-vaccination hSBA titer ≥1:4, an increase in hSBA titer of at least four times the pre-vaccination titer.
Time Frame: Day 29 (1 month post vaccination)
Population: Analysis was done on the Full Analysis Set (FAS), ie, all subjects in the exposed population who provided at least one evaluable serum sample whose assay result is available for at least one serogroup.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- 2 - 10 Years: Subjects between 2 and 10 years of age who received one injection of MenACWY -CRM vaccine on day 1.
- 11 - 18 Years: Subjects between 11 and 18 years of age who received one injection of MenACWY -CRM vaccine on day 1.
- 19 - 75 Years: Subjects between 19 and 75 years of age who received one injection of MenACWY -CRM vaccine on day 1.
- Overall (≥2 Years): Subjects between 2 and 75 years of age who received one injection of MenACWY -CRM vaccine on day 1.
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 59 | 58 | 177
Percentages of subjects | 75 [62 to 85] | 76 [63 to 86] | 66 [52 to 78] | 72 [65 to 79]

2. Primary Outcome: Percentages of Subjects With Human Serum Bactericidal Assay (hSBA) Seroresponse Against N.Meningitidis Serogroup C
Description: The immunogenicity of a single injection of MenACWY-CRM vaccine is assessed in terms of percentage of subjects with hSBA seroresponse directed against N.meningitidis serogroup C.
Time Frame: Day 29 (1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 58 | 59 | 58 | 175
Percentages of subjects | 84 [73 to 93] | 90 [79 to 96] | 90 [79 to 96] | 88 [82 to 92]

3. Primary Outcome: Percentages of Subjects With Human Serum Bactericidal Assay (hSBA) Seroresponse Against N.Meningitidis Serogroup W.
Description: The immunogenicity of a single injection of MenACWY-CRM vaccine is assessed in terms of percentage of subjects with hSBA seroresponse directed against N.meningitidis serogroup W.
Time Frame: Day 29 (1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 59 | 57 | 176
Percentages of subjects | 58 [45 to 71] | 51 [37 to 64] | 54 [41 to 68] | 55 [47 to 62]

4. Primary Outcome: Percentages of Subjects With Human Serum Bactericidal Assay (hSBA) Seroresponse Against N.Meningitidis Serogroup Y.
Description: The immunogenicity of a single injection of MenACWY-CRM vaccine is assessed in terms of percentage of subjects with hSBA seroresponse directed against N.meningitidis serogroup Y.
Time Frame: Day 29 (1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 58 | 59 | 57 | 174
Percentages of subjects | 69 [55 to 80] | 69 [56 to 81] | 75 [62 to 86] | 71 [64 to 78]

5. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup A at Day 1.
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup A at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 59 | 60 | 179
Percentage of subjects | 0 [0 to 6] | 2 [0 to 9] | 2 [0 to 9] | 1 [0 to 4]

6. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup A at Day 29.
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup A at day 29.
Time Frame: Day 29 (ie, 1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 58 | 178
Percentages of subjects | 75 [62 to 85] | 77 [64 to 87] | 66 [52 to 78] | 72 [65 to 79]

7. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup C at Day 1.
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup C at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 58 | 59 | 60 | 177
Percentages of subjects | 14 [6 to 25] | 24 [14 to 37] | 25 [15 to 38] | 21 [15 to 28]

8. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup C at Day 29.
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup C at day 29.
Time Frame: Day 29 (ie, 1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 58 | 178
Percentages of subjects | 92 [82 to 97] | 97 [88 to 100] | 97 [88 to 100] | 95 [91 to 98]

9. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup W at Day 1.
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup W at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 59 | 59 | 178
Percentages of subjects | 52 [38 to 65] | 63 [49 to 75] | 59 [46 to 72] | 58 [50 to 65]

10. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup W at Day 29.
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup W.
Time Frame: Day 29
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 58 | 178
Percentage of subjects | 95 [86 to 99] | 95 [86 to 99] | 93 [83 to 98] | 94 [90 to 97]

11. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup Y at Day 1
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup Y at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 59 | 59 | 59 | 177
Percentages of subjects | 22 [12 to 35] | 53 [39 to 66] | 53 [39 to 66] | 42 [35 to 50]

12. Secondary Outcome: Percentages of Subjects With hSBA ≥1:8 Directed Against N.Meningitidis Serogroup Y at Day 29
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by the percentage of subjects aged 2 through 75 with hSBA titer ≥ 1:8, directed against N. meningitidis serogroup Y at day 29.
Time Frame: Day 29 (ie, 1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 59 | 60 | 58 | 177
Percentages of subjects | 83 [71 to 92] | 95 [86 to 99] | 93 [83 to 98] | 90 [85 to 94]

13. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Directed Against N.Meningitidis Serogroup A at Day 1
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup A at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 59 | 60 | 179
Titer | 2.08 [1.97 to 2.20] | 2.05 [1.95 to 2.16] | 2.07 [1.93 to 2.21] | 2.07 [2.00 to 2.14]

14. Secondary Outcome: hSBA GMTs Directed Against N.Meningitidis Serogroup A at Day 29
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup A at day 29.
Time Frame: Day 29 ( ie, 1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 58 | 178
Titer | 30 [19 to 47] | 50 [30 to 84] | 29 [16 to 51] | 35 [26 to 47]

15. Secondary Outcome: hSBA GMTs Directed Against N.Meningitidis Serogroups C at Day 1
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup C at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 58 | 59 | 60 | 177
Titer | 2.88 [2.26 to 3.65] | 4.01 [3.00 to 5.35] | 4.14 [3.12 to 5.49] | 3.63 [3.11 to 4.25]

16. Secondary Outcome: hSBA GMTs Directed Against N.Meningitidis Serogroups C at Day 29
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup C at day 29.
Time Frame: Day 29 (ie, 1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 58 | 178
Titer | 67 [44 to 101] | 191 [117 to 310] | 287 [191 to 431] | 153 [117 to 199]

17. Secondary Outcome: hSBA GMTs Directed Against N.Meningitidis Serogroup W at Day 1
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup W at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 59 | 59 | 178
Titer | 9.27 [6.33 to 14] | 14 [9.13 to 20] | 12 [7.70 to 17] | 11 [9.05 to 14]

18. Secondary Outcome: hSBA GMTs Directed Against N.Meningitidis Serogroup W at Day 29
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup W at day 29.
Time Frame: Day 29 (ie, 1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 58 | 178
Titer | 60 [44 to 81] | 75 [54 to 105] | 116 [71 to 187] | 80 [64 to 100]

19. Secondary Outcome: hSBA GMTs Directed Against N.Meningitidis Serogroup Y at Day 1
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup Y at day 1.
Time Frame: Day 1
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 59 | 59 | 59 | 177
Titer | 3.59 [2.75 to 4.70] | 7.87 [5.48 to 11] | 8.69 [5.98 to 13] | 6.26 [5.13 to 7.65]

20. Secondary Outcome: hSBA GMTs Directed Against N.Meningitidis Serogroup Y at Day 29
Description: To assess the immunogenicity of a single injection of MenACWY-CRM vaccine as measured by hSBA GMTs directed against N. meningitidis serogroup Y at day 29.
Time Frame: Day 29 (ie, 1 month post vaccination)
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 59 | 60 | 58 | 177
Titer | 45 [29 to 69] | 105 [72 to 155] | 173 [97 to 309] | 93 [70 to 123]

21. Secondary Outcome: Number of Subjects Who Reported Any Solicited Local and Systemic Reactions Post Vaccination
Description: The safety of one dose of MenACWY - CRM was assessed in terms of the number of subjects reporting any solicited local and systemic reactions.
Time Frame: From day 1 to Day 7 post vaccination
Population: The analysis was performed on the safety analysis set, ie, all subjects in the exposed population who provided any post-baseline safety data.
Measure: Number; unit: Participants
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 60 | 180
Participants
  INJECTION SITE REACTIONS | 5 | 17 | 5 | 27
  SYSTEMIC REACTIONS | 3 | 7 | 9 | 19

22. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Reactions Post Vaccination
Description: The safety of one dose of MenACWY - CRM was assessed in terms of the number of subjects reporting solicited local and systemic reactions.
Time Frame: From day 1 to Day 7 post vaccination
Population: The analysis was performed on the safety analysis set.
Measure: Number; unit: Participants
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 60 | 180
Participants
  ANALGESIC ANTIPYRETIC | 2 | 5 | 2 | 9
  Body Temperature >=40C | 0 | 0 | 0 | 0
  ERYTHEMA (mm) | 0 | 0 | 0 | 0
  INDURATION (mm) | 0 | 0 | 0 | 0
  PAIN | 4 | 17 | 5 | 26
  TENDERNESS | 1 | 0 | 0 | 1
  ARTHRALGIA | 1 | 1 | 0 | 2
  BODY TEMPERATURE >=38C | 1 | 1 | 1 | 3
  CHANGE IN EATING HABITS | 0 | 0 | 0 | 0
  CHILLS | 0 | 4 | 2 | 6
  DIARRHEA | 0 | 0 | 0 | 0
  HEADACHE | 2 | 5 | 7 | 14
  IRRITABILITY | 0 | 0 | 0 | 0
  MALAISE | 2 | 2 | 2 | 6
  MYALGIA | 1 | 0 | 2 | 3
  NAUSEA | 0 | 1 | 1 | 2
  RASH | 0 | 0 | 0 | 0
  SLEEPINESS | 0 | 0 | 0 | 0
  VOMITING | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: The safety of one dose of MenACWY -CRM was assessed in terms of the number of subjects reporting unsolicited adverse events. All AEs were recorded from day 1 to day 7; SAE, medically attended AEs and AEs Leading to premature withdrawal were recorded throughout the entire study period.
Time Frame: Day 1 through day 29
Population: The analysis was performed on the safety analysis dataset.
Measure: Number; unit: participants
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Number analyzed (Participants) | 60 | 60 | 60 | 180
participants
  Any Unsolicited AE | 9 | 6 | 4 | 19
  Any SAE | 0 | 0 | 1 | 0
  Medically Attended AEs | 8 | 5 | 4 | 17
  AEs Leading to premature withdrawal | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 29 post vaccination.
Description: Any solicited and unsolicited adverse events were collected from 30 minutes post vaccination up to 7 days. Serious Adverse Events (SAE), medically attended AEs, AEs leading to withdrawal from the study were collected from day 1 through day 29.
Arm/Group | 2 - 10 Years | 11 - 18 Years | 19 - 75 Years | Overall (≥2 Years)
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 1/60 | 1/180
Other Adverse Events (participants affected / at risk) | 10/60 | 21/60 | 10/60 | 41/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 - 10 Years (N=60) | 11 - 18 Years (N=60) | 19 - 75 Years (N=60) | Overall (≥2 Years) (N=180)
PYREXIA (General disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 - 10 Years (N=60) | 11 - 18 Years (N=60) | 19 - 75 Years (N=60) | Overall (≥2 Years) (N=180)
CHILLS (General disorders) | 0 | 4 | 2 | 6
INJECTION SITE PAIN (General disorders) | 5 | 17 | 5 | 27
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 1 | 0 | 5
HEADACHE (Nervous system disorders) | 2 | 5 | 7 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less